CLINICAL TRIAL: NCT05854459
Title: Effects of High-intensity Interval Training With an Eccentric Hamstring Exercise Program in Futsal Players
Brief Title: HIIT With an Eccentric Hamstring Exercise Program in Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IE1541414
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT and Nordic Curl exercise group (Experimental): The participants will perform a weekly 50 minutes session for four weeks.
  Interventions: Other: HIIT and Nordic Curl exercise program
- HIIT-only group (Active Comparator): The participants will perform a weekly 40 minutes session for four weeks.
  Interventions: Other: HIIT-only program

INTERVENTIONS:
Other: HIIT and Nordic Curl exercise program — The training program in the HIIT+NC group was divided into the following parts: i) warm-up (10 minutes); ii) HIIT (25 minutes) consisting of a circuit of eight exercises; iii) Nordic curl exercise (10 mintues); and iv) stretching.
  Arms: HIIT and Nordic Curl exercise group
Other: HIIT-only program — The HIIT group performed the same exercises in the warm-up, HIIT and stretching sections as the HIIT+NC group, however, they did not perform the NC eccentric exercises.
  Arms: HIIT-only group

SUMMARY:
Physiotherapy protocols based on high-intensity interval training (HIIT) or eccentric hamstring exercises like Nordic Curl (NC) have been scarcely studied in futsal players. The hypothesis of this study is that a HIIT combined with an NC exercise program is more effective than a HIIT-only program in improving physical and functional characteristics in futsal players.

DETAILED DESCRIPTION:
The objective of this study was to compare the effectiveness of a HIIT combined with an NC exercise program versus a HIIT-only program in futsal players. Therefore, a randomized controlled trial will be carried out. Futsal players will be divided into 1) HIIT+NC group and 2) HIIT group. The HIIT+NC group will perform a HIIT circuit combined with 3 sets of 10 NC repetitions for 4 weeks, while the HIIT group will perform the same protocol without NC exercise. BMI, intermittent work performance, vertical jump performance without and with arms, isometric strength of quadriceps and hamstrings, and the isometric H/Q ratio, will be assessed before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Futsal players, over 18 years of age.

Exclusion Criteria:

* Those who had a medical condition that prevented them from performing any of the evaluations.
* Those who declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Intermittent work performance | Baseline
  Intermittent work performance will be assessed with the 30x15 Intermittence Test (30x15IFT). The speed of the test will be recorded in km/h. The higher the speed achieved, the better work performance.
Intermittent work performance | After the intervention (4 weeks)
  Intermittent work performance will be assessed with the 30x15 Intermittence Test (30x15IFT). The speed of the test will be recorded in km/h. The higher the speed achieved, the better the work performance.

SECONDARY OUTCOMES:
Vertical jump performance without arm impulse | Baseline
  Vertical jump performance without arm impulse will be measured with the Counter Movement Jumping Test (CMJ). The jump height was calculated using the My Jump 2 program (My Jump Lab, Madrid, Spain) in cm. The higher the height achieved, the better the vertical jump performance.
Vertical jump performance without arm impulse | After the intervention (4 weeks)
  Vertical jump performance without arm impulse will be measured with the Counter Movement Jumping Test (CMJ). The jump height was calculated using the My Jump 2 program (My Jump Lab, Madrid, Spain) in cm. The higher the height achieved, the better the vertical jump performance.
Vertical jump performance with arm impulse | Baseline
  Vertical jump performance with arm impulse will be measured with the Counter Movement Jumping Test (CMJ). The jump height was calculated using the My Jump 2 program (My Jump Lab, Madrid, Spain) in cm. The higher the height achieved, the better the vertical jump performance.
Vertical jump performance with arm impulse | After the intervention (4 weeks)
  Vertical jump performance with arm impulse will be measured with the Counter Movement Jumping Test (CMJ). The jump height was calculated using the My Jump 2 program (My Jump Lab, Madrid, Spain) in cm. The higher the height achieved, the better the vertical jump performance.
Maximal quadriceps isometric strength | Baseline
  Maximal quadriceps isometric strength will be measured using the Adapted Quadriceps Sphygmomanometer Test in mmHg. The higher the pressure (mmHg) achieved, the better the quadriceps isometric strength.
Maximal quadriceps isometric strength | After the intervention (4 weeks)
  Maximal quadriceps isometric strength will be measured using the Adapted Quadriceps Sphygmomanometer Test in mmHg. The higher the pressure (mmHg) achieved, the better the quadriceps isometric strength.
Maximal hamstrings isometric strength | Baseline
  Maximal hamstrings isometric strength will be measured using the Adapted Hamstrings Sphygmomanometer Test in mmHg. The higher the pressure (mmHg) achieved, the better the hamstrings isometric strength.
Maximal hamstrings isometric strength | After the intervention (4 weeks)
  Maximal hamstrings isometric strength will be measured using the Adapted Hamstrings Sphygmomanometer Test in mmHg. The higher the pressure (mmHg) achieved, the better the hamstrings isometric strength.
Isometric hamstrings/quadriceps ratio | Baseline
  Isometric hamstrings/quadriceps (H/Q) ratio will be calculated by dividing the values obtained previously in the maximum isometric strength test of the hamstrings by those obtained in the quadriceps test. The value closer to 1, the greater the balance between the hamstrings and quadriceps muscles.
Isometric hamstrings/quadriceps ratio | After the intervention (4 weeks)
  Isometric hamstrings/quadriceps (H/Q) ratio will be calculated by dividing the values obtained previously in the maximum isometric strength test of the hamstrings by those obtained in the quadriceps test. The value closer to 1, the greater the balance between the hamstrings and quadriceps muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marqués Sulé, Dr, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos FS, Borszcz FK, Flores LJF, Barazetti LK, Teixeira AS, Hartmann Nunes RF, Guglielmo LGA. HIIT Models in Addition to Training Load and Heart Rate Variability Are Related With Physiological and Performance Adaptations After 10-Weeks of Training in Young Futsal Players. Front Psychol. 2021 Jan 22;12:636153. doi: 10.3389/fpsyg.2021.636153. eCollection 2021. PMID 33551944
- [Background] Krommes K, Petersen J, Nielsen MB, Aagaard P, Holmich P, Thorborg K. Sprint and jump performance in elite male soccer players following a 10-week Nordic Hamstring exercise Protocol: a randomised pilot study. BMC Res Notes. 2017 Dec 4;10(1):669. doi: 10.1186/s13104-017-2986-x. PMID 29202784